CLINICAL TRIAL: NCT04058223
Title: Taipei Medical University Shuang-Ho Hospital
Brief Title: Comparison of the Short-term Outcomes of Using DST and PPH Staplers in the Treatment of Grade III and IV Hemorrhoids
Status: Completed | Type: Observational
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Tungcheng Chang, Chief of colorectal surgery, Taipei Medical University Shuang Ho Hospital
Other Study IDs: N201808042
Record Dates: First submitted 2019-08-14; First posted 2019-08-15 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Bleeding; Stricture
MeSH Terms: conditions — Hemorrhage; Constriction, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — After the surgery, the ring of the excised anorectal mucosa was cut open and flattened on a surgical towel as shown in Figure 2. The presence of muscle in the specimen was confirmed grossly and photographed. The entire surface area of the mucosa, muscle and the muscle/mucosa ratio were measured using the ImageJ software (National Institutes of Health, Bethesda, MD, USA).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PPH/DST: Patients underwent hemorrhoidopexy by PPH or DST stapler.
  Interventions: Device: Hemorrhoidopexy

INTERVENTIONS:
Device: Hemorrhoidopexy — stapled hemorrhoidopexy

SUMMARY:
The hemorrhoidal disease affects approximately 4.4%-36% of the general population, and it has been estimated that >50% of the population aged >50 years experiences hemorrhoidal problems . Traditional hemorrhoidectomy, including Milligan-Morgan, Ferguson, and Whitehead procedures , are known to cause significant postoperative pain and discomfort and result in a poor quality of life after operation. Since the first introduction of the novel procedure hemorrhoidopexy by Longo in 1998, it has been considered as a safe procedure causing less postoperative pain and resulting in earlier recovery; furthermore, the patients are able to resume their normal daily life and work. The PPH stapler (Ethicon Endo-Surgery, Inc. Cincinnati, OH, USA) was also first introduced in 1998 as a device to perform this procedure. Subsequently, a new device, the DST stapler (Covidien, Mansfield, MA, USA), was introduced in 2008 with some structural differences, including a detachable anvil, three anchor points over different levels, a larger case, and different agraffe sizes.

However, the majority of current studies have been focusing on the use of PPH stapler for hemorrhoidopexy, and comparison with the DST stapler has been rarely discussed. One randomized controlled trial that compared between the PPH stapler and the DST stapler reported that the DST stapler demonstrated a better hemostatic ability and allowed the resection of a larger area of mucosal prolapse; however, that trial focused only on bleeding among the postoperative complications. Currently, only a limited number of studies have compared these two devices in terms of pain, complications, and anorectal stricture incidence rate. The present investigation is a matched cohort-control study aimed to compare the postoperative short-term outcomes among patients with grade III and IV hemorrhoids who were treated with either the PPH or the DST stapler. The specimen surface area and the relationships with complications were also analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Grade III and grade IV hemorrhoid

Exclusion Criteria:

* Anal fistula, rectal polyo\p

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with grade III and IV hemorrhoid underwent stapled hemorrhoidopexy
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
Complication | 3 months
  Post-OP bleeding, urinary retention, anaorectal stricture, PPH syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Tung-Cheng Chang, MD, PHD, Study Director — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Taipei Medical University Shuang-Ho Hospital, New Taipei City, Taiwan